CLINICAL TRIAL: NCT06589232
Title: Threshold Dose Distribution for Pistachio Allergy in Children
Brief Title: Threshold Dose Distribution for Pistachio Allergy
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Amandine DIVARET-CHAUVEAU, Principal investigator, Central Hospital, Nancy, France
Other Study IDs: 2024PI051
Record Dates: First submitted 2024-04-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Allergy; Food Allergy
MeSH Terms: conditions — Hypersensitivity; Food Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Food allergy: Threshold dose to pistachio
  Interventions: Other: Food allergy

INTERVENTIONS:
Other: Food allergy — Threshold dose to pistachio

SUMMARY:
The main objective of this study is to describe the distribution of reactogenic thresholds for pistachio. The secondary objectives are to 1) describe the clinical severity of allergic reactions to pistachio in an oral challenge test, 2) compare the reactogenic thresholds of pistachio and cashew nut on matched data and 3) evaluate predictive factors of a low reactogenic threshold

DETAILED DESCRIPTION:
Nuts, including almonds, walnuts, cashews, pistachio and hazelnut, are among the food allergens most frequently involved in food allergies in children with an estimated prevalence. between 0.05 and 4.9%.

According to data from the Allergo-Vigilance Network, peanuts and the group of nuts, led by cashews, are alone responsible for 51.4% of food anaphylaxis in children.

The pistachio belongs to the same botanical family as the cashew nut (Anacardiumouest) and the mango (Mangifera indica): the anacardiaceae. Botanically, pistachio and cashew are closely related and can both be responsible for moderate to severe immediate allergic reactions. Furthermore, in a previous publication by the team, co-sensitization to pistachio was observed in 98% of children allergic to cashew nuts with only 34% confirmed allergic to pistachio.

In the case of allergy to both anacardiaceae, in a small number of patients, the investigators reported a reactogenic threshold for pistachio greater than or equal to that for cashew nuts.

To our knowledge, there is currently only one study that has evaluated the reactogenic threshold for pistachio, compared to other nuts.

ELIGIBILITY:
Inclusion Criteria:

* Patients under 18 years of age who had a positive pistachio challenge test between January 2021 and December 2023, in the pediatric allergology unit of the Nancy CHRU.

Exclusion Criteria:

* Patients who had a questionable oral pistachio provocation test.
* Patients who had a negative pistachio oral provocation test.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients under 18 years of age who had a positive pistachio challenge test between January 2021 and December 2023, in the pediatric allergology unit of the Nancy CHRU
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-09 (Actual)

PRIMARY OUTCOMES:
Threshold dose to pistachio | in the 4 hours of monitoring
  in mg of protein

SECONDARY OUTCOMES:
Threshold dose to cashew | in the 4 hours of monitoring
  in mg of proteins
Severity of the reaction during a positive pistachio oral provocation test | in the 4 hours of monitoring
  defined by the COFAR (Consortium for Food Allergy Research) classification, from 1 to 5 and 1 is for mild symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Amandine DIVARET-CHAUVEAU, Principal Investigator — Centre hospitalo-universitaire de Nancy
Locations (1):
- Centre Hospitalo-Universitaire de Nancy, Vandœuvre-lès-Nancy, France, France

IPD SHARING:
Plan to Share IPD: No